CLINICAL TRIAL: NCT01193153
Title: A Randomized, Double-Blind, Placebo-Controlled, Parellel-Group Study of Paliperidone Palmitate Evaluating Time to Relapse in Subjects With Schizoaffective Disorder
Brief Title: A Study to Evaluate the Efficacy of Paliperidone Palmitate in the Prevention of Relapse of the Symptoms of Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR016618; R092670SCA3004 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Schizoaffective Disorder
Keywords: schizoaffective disorder; paliperidone palmitate; INVEGA SUSTENNA; schizoaffective disorder relapse prevention
MeSH Terms: conditions — Psychotic Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): paliperidone palmitate 78 117 156 234 mg (50 75 100 or 150 mg eq.) monthly by i.m. injection for 15 months
  Interventions: Drug: paliperidone palmitate
- 002 (Placebo Comparator): Placebo monthly by i.m. injection for 15 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — monthly by i.m. injection for 15 months
  Arms: 002
Drug: paliperidone palmitate — 78, 117, 156, 234 mg (50, 75, 100, or 150 mg eq.) monthly by i.m. injection for 15 months
  Arms: 001

SUMMARY:
This study will evaluate the efficacy of paliperidone palmitate compared with placebo in the delay of relapse of the symptoms of schizoaffective disorder. This study will also assess the safety and tolerability of paliperidone palmitate in patients with schizoaffective disorder.

DETAILED DESCRIPTION:
Schizoaffective disorder is a chronic illness and generally requires life-long treatment. To date however, no medication has been evaluated in the maintenance treatment of schizoaffective disorder. This is a randomized (study drug assigned by chance), double-blind (neither physician nor patient knows the name of the assigned drug), placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of paliperidone palmitate, as monotherapy or as an adjunct to mood stabilizers or antidepressants, relative to placebo in delaying the time to relapse in patients with schizoaffective disorder. This study explores the use of paliperidone palmitate either as monotherapy or as an adjunct to mood stabilizers or antidepressants (MS/AD) because both treatment approaches are commonly used in the clinical management of schizoaffective disorder. Patients with acute symptoms of schizoaffective disorder will be enrolled. The study will consist of 4 periods: an up to 7 days screening/tolerability period, a 13-week open-label flexible dose lead-in period, a 12-week open-label fixed dose stabilization period, and a 15 months double-blind relapse prevention period. Patients without previous exposure to paliperidone ER (Invega), paliperidone palmitate (Invega Sustenna), risperidone, or RISPERDAL CONSTA will be given 4 to 6 days of paliperidone ER 6mg/day for tolerability testing. Patients can continue their current antipsychotic regimen through Day -1 (the day before the start of the study period). During the open-label periods, all patients will be treated with paliperidone palmitate. An initial loading dose of 234 mg (150 mg eq.) of paliperidone palmitate will be given by deltoid injection followed by 156 mg (100 mg eq.) deltoid injection on Day 8. Starting on Day 36, injections may be administered in either the deltoid muscle or the gluteal muscle. Doses at Days 36, 64 and 92 may be increased or decreased within the range of 78 mg (50 mg eq.) and 234 mg (150 mg. eq.) as clinically indicated. Dose will be fixed (at Day 92 dose) during the 12-week stabilization period. Patients who meet pre-determined stabilization criteria will be eligible to enter the double-blind relapse prevention period and will be randomly assigned to either receive paliperidone palmitate (at the Day 92 dose) or placebo treatment. Patients will have intramuscular (i.m.) study drug injection and efficay and saftety evaluations performed every 4 weeks throughout the study. Efficacy will be evaluated during the study using a relapse assessment, the Positive and Negative Symptom Scale (PANSS), the Clinical Global Impression of Severity for Schizoaffective Disorder (CGI-S-SCA), the Personal and Social Performance Scale (PSP), the Young Mania Rating Scale (YMRS), and the Hamilton Rating Scale for Depression (HAM-D). Safety will be assessed throughout the study by monitoring of adverse events, clinical laboratory tests, electrocardiograms (ECGs), vital sign measurements (temperature, pulse, and blood pressure), weight, and the monitoring of extrapyramidal symptoms using the Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A). Suicidality will be assessed by the Columbia Suicide Severity Rating Scale (C-SSRS). A 10 milliliter pharmacogenomic blood sample (sample for DNA research) will be collected from patients who give separate written informed consent for this part of the study. Participation in pharmacogenomic research is optional. Blood samples will be taken from patients being treated with lithium or valproate for the measurement of blood lithium or valproate levels. Approximately 52 mL (31 mL for patients who are not receiving lithium or valproate) of whole blood will be collected during the study. All patients will receive paliperidone palmitate 78, 117, 156, 234 mg (50, 75, 100, or 150 mg eq.) monthly by i.m. injection for the the first 25 weeks of the study (open-label periods). During the 15-month double-blind relapse prevention period, one half of the patients will be randomized to paliperidone palmitate treatment (50, 75, 100, or 150 mg eq. monthly i.m. injection) and the other half of the patients will be randomized to monthly placebo injection.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizoaffective disorder
* Experiencing an acute exacerbation of psychotic symptoms
* A score of >=4 on at least 3 of the following 7 PANSS items: Delusions (P1), Hallucinatory behavior (P3), Excitement (P4), Hostility (P7), Tension (G4), Uncooperativeness (G8), and Poor Impulse Control (G14)
* A score of >=16 on YMRS and/or a score of >=16 on the HAM-D-21
* Healthy based on physical examinations, electrocardiogram (ECG), laboratory tests, medical history, and vital signs measurements

Exclusion Criteria:

* A primary active mental illness diagnosis other than schizoaffective disorder
* Have attempted suicide within 12 months or are at imminent risk of suicide or violent behavior
* Subjects with first episode of psychosis
* Received electroconvulsive therapy in the past 3 months
* History of hypersensitivity to or intolerance of paliperidone, risperidone, or 20% Intralipid (placebo)
* Received long-acting antipsychotic medication within 2 injection cycles
* Received therapy with clozapine within 3 months
* A history of neuroleptic malignant syndrome
* Previous history of lack of response to antipsychotic medication
* Subjects receiving therapy with antidepressants or mood stabilizers that has been initiated and/or changed in dose <30 days prior to screening
* Receiving therapy with carbamazepine
* Receiving therapy with monoamine oxidase inhibitors
* Pregnant, breast-feeding, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (80):
- United States (28):
  - Garden Grove, California
  - Oakland, California
  - Oceanside, California
  - Pico Rivera, California
  - Riverside, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Hollywood, Florida
  - Maitland, Florida
  - North Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Schamburg, Illinois
  - Wichita, Kansas
  - Flowood, Mississippi
  - Creve Coeur, Missouri
  - Cedarhurst, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - Irving, Texas
  - San Antonio, Texas
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
- India (13):
  - Ahmedabad
  - Aurangabad
  - Chennai
  - Jaipur
  - Lucknow Gpo
  - Mangalore
  - Mysore
  - Nashik
  - Pune
  - Uttar Pradesh
  - Vadadora
  - Varanasi
  - Vijaywada
- Malaysia (6):
  - Alor Star
  - Ipoh
  - Kota Bharu
  - Kota Kinabalu
  - Kuala Lumpur
  - Tanjong Rambutan
- Philippines (4):
  - Cebu
  - Davao City
  - Iloilo City
  - Quezon City
- Romania (7):
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Oradea
  - Sibiu
  - Timișoara
- South Africa (7):
  - Cape Town
  - Centurion Gauteng
  - Durban
  - George
  - Johannesburg
  - Pretoria
  - Tyger Valley
- Ukraine (11):
  - Dnipropetrovsk
  - Donetsk
  - Hlevakha
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Poltava
  - Simferopol
  - Uzhhorod
  - Village Stepanovka Kherson
  - Vinnitsa

REFERENCES:
- [Derived] Alphs L, Fu DJ, Turkoz I. Paliperidone for the treatment of schizoaffective disorder. Expert Opin Pharmacother. 2016;17(6):871-83. doi: 10.1517/14656566.2016.1161029. Epub 2016 Mar 24. PMID 26934062
- [Derived] Fu DJ, Turkoz I, Simonson RB, Walling DP, Schooler NR, Lindenmayer JP, Canuso CM, Alphs L. Paliperidone palmitate once-monthly reduces risk of relapse of psychotic, depressive, and manic symptoms and maintains functioning in a double-blind, randomized study of schizoaffective disorder. J Clin Psychiatry. 2015 Mar;76(3):253-62. doi: 10.4088/JCP.14m09416. PMID 25562685

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants without previous exposure to paliperidone extended-release (ER) (Invega), or risperidone, received paliperidone ER 6 milligram (mg)/day for 4 to 6 days (during Screening) to test oral tolerability. Only participants, who had ability to tolerate the drug, as judged by treating physician, were eligible for enrollment in the study.
Groups:
- Paliperidone Palmitate: Open Label (OL) Lead-in (13 weeks): 234 milligram (mg) injection on Day 1, 156 mg on Day 8, flexible dose between 78-234 mg on Days 36, 64, and 92. Participants who met criteria: Positive and Negative Syndrome Scale (PANSS) total score less than or equal to (<=) 70, and Young Mania Rating Scale [YMRS] and Hamilton Rating Scale for Depression [HAM-D-21] <=12 at the end of open label lead-in period entered stabilization period. OL Stabilization (12 weeks): Same dose as Day 92 in OL lead in period, on Day 120 once every 4 weeks. Participants who completed stabilization period and maintained stabilization criteria throughout 12 weeks entered double- bind (DB) relapse prevention period. DB Relapse prevention period (15 months): Same dose as Day 92 once every 4 weeks until one of the following occurred: met the prospectively defined relapse criteria; discontinued treatment for a reason other than relapse; withdrew consent; lost to follow-up; completed 15 months of double-blind treatment.
- Placebo: Participants did not receive placebo during OL lead in period and OL stabilization period. Participants received matching placebo injections of 20 percent Intralipid (200 milligram per milliliter [mg/mL]) emulsion, once every 4 weeks during double-blind relapse prevention period.
Period: Open-label Lead in Period
Arm/Group | Paliperidone Palmitate | Placebo
Started | 667 | 0
Completed | 432 | 0
Not Completed | 235 | 0
Not completed — Lost to Follow-up | 32 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 69 | 0
Not completed — > 6 Weeks Between 2 Study Drug | 4 | 0
Not completed — Other | 14 | 0
Not completed — Subject Failed Stabilization Criteria | 47 | 0
Not completed — Adverse Event | 41 | 0
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 26 | 0
Period: Open-label Stabilization Period
Arm/Group | Paliperidone Palmitate | Placebo
Started | 432 | 0
Completed | 334 | 0
Not Completed | 98 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 10 | 0
Not completed — Lack of Efficacy | 5 | 0
Not completed — Withdrawal by Subject | 29 | 0
Not completed — Subject Failed Stabilization Criteria | 35 | 0
Not completed — Other | 8 | 0
Period: Double Blind Relapse Prevention Period
Arm/Group | Paliperidone Palmitate | Placebo
Started | 164 | 170
Completed | 100 | 65
Not Completed | 64 | 105
Not completed — Other | 2 | 3
Not completed — Adverse Event | 12 | 3
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 2 | 9
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 19 | 30
Not completed — Experienced Relapse | 25 | 57
Not completed — > 6 Weeks Between 2 Study Drug | 1 | 3

BASELINE CHARACTERISTICS:
Population: Open-label (OL) intent-to-treat (ITT) analysis set included all participants who received at least 1 injection of open-label study drug.
Groups:
- Entire Study Population: Included all participants who received at least 1 dose of paliperidone palmitate in open-label lead in period.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 667
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310
  Male | 357

OUTCOME MEASURES:

1. Primary Outcome: Double-blind: Percentage of Participants Who Experienced Relapse
Description: Relapse was defined as first occurrence of any 1 of following:psychiatric hospitalization due to worsening symptoms; any intervention employed to avert imminent hospitalization due to worsening symptoms or need for additional antipsychotic,antidepressants/mood stabilizing medication; deliberate self-injury,suicidal/homicidal ideation that is clinically significant as determined by investigator,or violent behavior resulting in clinically significant injury to another person or property damage; worsening of any 1 or more of 8 selected positive and negative syndrome scale(PANSS) items to a score of greater than or equal to (>= 6) after randomization(if the score for the corresponding item was less than or equal to [<=] 4 at randomization); worsening of certain other measures in specific ways at 2 consecutive visits. Relapse by subgroup of participants on monotherapy,adjunctive therapy to antidepressants/mood stabilizers,participants with psychotic symptoms/mood symptoms was examined.
Time Frame: Day 1 up to Month 15 of double blind relapse prevention period
Population: Double-blind(DB) Intent-to-Treat(ITT) analysis set included all randomly assigned participants who received at least 1 injection of DB study medication.'n' signifies participants who were evaluable for each specified category,for each arm.
Measure: Number; unit: percentage of participants
Groups:
- Paliperidone Palmitate: DB Relapse prevention period (15 months): Same dose as Day 92, once every 4 weeks, given as monotherapy and as an adjunct to mood stabilizers or antidepressants, until one of the following occurred: met the prospectively defined relapse criteria; discontinued treatment for a reason other than relapse; withdrew consent; lost to follow-up; completed 15 months of double-blind treatment.
- Placebo: Matching placebo injections of 20 percent Intralipid (200 milligram per milliliter [mg/mL]) emulsion, once every 4 weeks, given as monotherapy and as an adjunct to mood stabilizers or antidepressants.
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
percentage of participants
  All Participants (n=164, 170) | 15.2 [NA to NA] | 33.5 [NA to NA]
  Monotherapy subset (n=78, 73) | 11.5 | 32.9
  Adjunct therapy subset (n=86, 97) | 18.6 | 34.0
  Psychotic Symptoms (n=164, 170) | 12.8 | 31.2
  Mood Symptoms;Any Mood Symptoms (n=164, 170) | 11.0 | 28.2
  Mood Symptoms;Manic (n=164, 170) | 3.0 | 9.4
  Mood Symptoms;Depressive (n=164, 170) | 4.9 | 13.5
  Mood Symptoms; Mixed (n=164, 170) | 3.0 | 5.3
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Placebo; All participants: p-value was calculated using log-rank test; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 2.49, 95% CI 2-sided [1.55 to 3.99]
Statistical Analysis 2: Comparison: Paliperidone Palmitate vs Placebo; Monotherapy subset: Hazard ratio and corresponding p-value, and 95% Confidence Interval (CI) were calculated from Cox proportional hazard regression model; Test type: Superiority or Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 3.38, 95% CI 2-sided [1.57 to 7.28]
Statistical Analysis 3: Comparison: Paliperidone Palmitate vs Placebo; Adjunct therapy subset: Hazard ratio and corresponding p-value, and 95% CI were calculated from Cox proportional hazard regression model; Test type: Superiority or Other; p = 0.021, Regression, Cox; Hazard Ratio (HR) = 2.03, 95% CI 2-sided [1.11 to 3.68]
Statistical Analysis 4: Comparison: Paliperidone Palmitate vs Placebo; Psychotic Symptoms: Hazard ratio and corresponding p-value, and 95% CI were calculated from Cox proportional hazard regression model; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.82, 95% CI 2-sided [1.70 to 4.67]
Statistical Analysis 5: Comparison: Paliperidone Palmitate vs Placebo; Mood Symptoms (Any Mood Symptoms):Hazard ratio and corresponding p-value, and 95% CI were calculated from Cox proportional hazard regression model; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.93, 95% CI 2-sided [1.70 to 5.04]
Statistical Analysis 6: Comparison: Paliperidone Palmitate vs Placebo; Mood Symptoms (Manic): Hazard ratio and corresponding p-value, and 95% CI were calculated from Cox proportional hazard regression model; Test type: Superiority or Other; p = 0.012, Regression, Cox; Hazard Ratio (HR) = 3.62, 95% CI 2-sided [1.32 to 9.89]
Statistical Analysis 7: Comparison: Paliperidone Palmitate vs Placebo; Mood Symptoms (Depressive): Hazard ratio and corresponding p-value, and 95% CI were calculated from Cox proportional hazard regression model; Test type: Superiority or Other; p = 0.006, Regression, Cox; Hazard Ratio (HR) = 3.12, 95% CI 2-sided [1.39 to 6.98]
Statistical Analysis 8: Comparison: Paliperidone Palmitate vs Placebo; Mood Symptoms (Mixed): Hazard ratio and corresponding p-value, and 95% CI were calculated from Cox proportional hazard regression model; Test type: Superiority or Other; p = 0.238, Regression, Cox; Hazard Ratio (HR) = 1.93, 95% CI 2-sided [0.65 to 5.78]

2. Secondary Outcome: Double-blind: Change From Baseline in Personal and Social Performance (PSP) Total Score at Week 64 (Total Mixed Model Repeated Measures [MMRM] Analysis of Covariance [ANCOVA])
Description: The PSP scale was designed to assess the degree of dysfunction a participant exhibits during a month prior to any visit within 4 domains of behavior: a) socially useful activities, b) personal and social relationships, c) self-care, and d) disturbing and aggressive behavior, each rated on 6-point scale (1=absent to 6=very severe). Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning. A score lying between 71 and 100 indicated a good functioning; one between 31 and 70 indicated varying degrees of difficulty, and a score of <=30 indicated functioning so poor that participant required intensive supervision.
Time Frame: Baseline and Week 64 of double blind relapse prevention period
Population: DB ITT analysis set which included all randomly assigned participants who received at least one injection of double-blind study medication. 'n' signifies participants who were evaluable at each specified time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
Units on a scale
  Baseline (n=164, 170) | 72.8 (0.81) | 74.5 (0.81)
  Change at Week 64 (n=98, 65) | 2.0 (0.92) | -1.3 (1.03)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Placebo; The null hypothesis is that there is no difference in the mean of the PSP total score between the two treatment groups; Test type: Superiority or Other; p = 0.014, MMRM ANCOVA — P-value based on change from DB baseline in PSP score and was analyzed using mixed-model repeated measures analysis of covariance based on observed data; within-participant repeated measures were modeled using an unstructured covariance matrix; Least Square Mean Difference = 3.3, 95% CI 2-sided [0.68 to 5.95], Standard Error of Mean 1.33

3. Secondary Outcome: Open-label: Change From Baseline in Personal and Social Performance (PSP) Total Score at Endpoint
Description: as for outcome 2
Time Frame: Baseline and Endpoint (Week 13/LOCF) in Open-label (OL) Lead-in period, Endpoint (Week 25/LOCF) in open-label stabilization period
Population: OL ITT analysis set which included all randomly assigned participants who received at least one injection of open-label study medication. Last Observation Carried Forward (LOCF) method was used to impute missing values. 'n' signifies participants who were evaluable at each specified time point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Paliperidone Palmitate: Open Label (OL) Lead-in (13 weeks): 234 milligram (mg) injection on Day 1, 156 mg on Day 8, flexible dose between 78-234 mg on Days 36, 64, and 92, given as monotherapy and as an adjunct to mood stabilizers or antidepressants. Participants who met criteria: Positive and Negative Syndrome Scale (PANSS) total score less than or equal to (<=) 70, and Young Mania Rating Scale [YMRS] and Hamilton Rating Scale for Depression [HAM-D-21] <=12 at the end of open label lead-in period entered stabilization period. OL Stabilization (12 weeks): Same dose as Day 92 in OL lead in period, on Day 120 once every 4 weeks, given as monotherapy and as an adjunct to mood stabilizers or antidepressants.
- Placebo: Participants did not receive placebo during open-label lead in period and open-label stabilization period.
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 667 | 0
Units on a Scale
  OL Lead-in Period:Baseline (n=667) | 51.4 (11.02) |
  OL Lead-in Period:Change at Endpoint (n=622) | 12.6 (13.71) |
  OL Stabilization Period:Change at Endpoint (n=622) | 13.8 (14.92) |

4. Secondary Outcome: Double-blind: Change From Baseline in Personal and Social Performance (PSP) Total Score at Endpoint
Description: as for outcome 2
Time Frame: Baseline and Endpoint (Week 64/LOCF) in double-blind period
Population: DB ITT analysis set which included all randomly assigned participants who received at least one injection of double-blind study medication. LOCF method was used to impute missing values. 'n' signifies participants who were evaluable at each specified time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
Units on a Scale
  Double-blind: Baseline (n=164, 170) | 74.5 (0.81) | 72.8 (0.81)
  Double-blind: Change at Endpoint (n=161,168) | 0.5 (1.15) | -4.1 (1.13)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Change at Endpoint (Week 64/LOCF); Least Square Mean Difference = 4.5, 95% CI 2-sided [1.94 to 7.15]

5. Secondary Outcome: Double-blind: Number of Participants With Personal and Social Performance (PSP) Categorical Scores
Description: The PSP scale was designed to assess the degree of dysfunction a participant exhibits during a month prior to any visit within 4 domains of behavior: a) socially useful activities, b) personal and social relationships, c) self-care, and d) disturbing and aggressive behavior, each rated on 6-point scale (1=absent to 6=very severe). Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning. Number of participants in each specific category; good functioning (PSP total score >70), variable functioning (PSP total score between 31 and 70), and poor functioning (PSP total score <=30) were assessed.
Time Frame: Baseline and Endpoint (Week 64/LOCF) in DB period
Population: DB ITT analysis set which included all randomly assigned participants who received at least one injection of double-blind study medication. LOCF method was used to impute missing values.'n' signifies participants who were evaluable at each specified time point for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
participants
  Baseline: Poor (n=164, 170) | 0 | 0
  Baseline: Variable (n=164, 170) | 69 | 84
  Baseline: Good (n=164, 170) | 95 | 86
  Endpoint: Poor (n=161, 168) | 1 | 4
  Endpoint: Variable (n=161, 168) | 65 | 95
  Endpoint: Good (n=161, 168) | 95 | 69

6. Secondary Outcome: Open-label: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Endpoint
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline and Endpoint (Week 13/LOCF) in OL Lead-in period, Endpoint (Week 25/LOCF) in open-label stabilization period
Population: OL ITT analysis set which included all randomly assigned participants who received at least one injection of open-label study medication. LOCF method was used to impute missing values. 'n' signifies participants who were evaluable at each specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 667 | 0
Units on a scale
  OL Lead-in Period:Baseline (n=667) | 85.8 (12.76) |
  OL Lead-in Period:Change at Endpoint (n=653) | -21.8 (16.39) |
  OL Stabilization Period:Change at Endpoint (n=653) | -23.8 (18.30) |

7. Secondary Outcome: Double-blind: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Endpoint
Description: as for outcome 6
Time Frame: Baseline and Endpoint (Week 64/LOCF) in double-blind period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
Units on a scale
  Double-blind: Baseline (n=164, 170) | 51.1 (9.50) | 51.8 (9.47)
  Double-blind: Change at Endpoint (n=161, 168) | 0.5 (14.01) | 7.4 (18.53)

8. Secondary Outcome: Open-label: Change From Baseline in Hamilton Rating Scale for Depression (HAM-D-21) Total Score at Endpoint
Description: The HAM-D-21 is a 21-item, clinician-rated scale to evaluate depressed mood as well as the vegetative and cognitive symptoms of depression. The items are rated on a 5-point (0 to 4) scale. The 5-point scale items use a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A rating of 4 is usually reserved for extreme symptoms. The responses for all 21 items are summed to yield the HAM-D-21 total score that ranges from 0-63.
Time Frame: Baseline and Endpoint (Week 13/LOCF) in OL Lead-in period, Endpoint (Week 25/LOCF) in open-label stabilization period
Population: OL ITT analysis set which included all randomly assigned participants who received at least one injection of open-label study medication. LOCF method was used to impute missing values. n' signifies participants who were evaluable at each specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 667 | 0
Units on a scale
  OL Lead-in Period:Baseline (n=667) | 20.4 (7.81) |
  OL Lead-in Period:Change at Endpoint (n=653) | -9.7 (8.53) |
  OL Stabilization Period:Change at Endpoint (n=653) | -9.9 (9.08) |

9. Secondary Outcome: Double-blind: Change From Baseline in Hamilton Rating Scale for Depression (HAM-D-21) Total Score at Endpoint
Description: as for outcome 8
Time Frame: Baseline and Endpoint (Week 64/LOCF) in double-blind period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
Units on a scale
  Double-blind: Baseline (n=164, 170) | 5.7 (3.24) | 5.6 (3.32)
  Double-blind: Change at Endpoint (n=161, 168) | 0.8 (5.40) | 3.4 (7.42)

10. Secondary Outcome: Open-label: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Endpoint
Description: The YMRS was designed to measure the severity of manic symptoms, to gauge the effect of treatment on mania severity, and to detect a return of manic symptoms (for example relapse or recurrence). YMRS is a checklist of 11 items that are ranked on a scale of 0 to 4 or 0 to 8. Seven of the items (elevated mood, increased motor activity, sexual interest, sleep, language-thought disorder, appearance, and insight) are ranked 0 to 4 and have descriptors associated with each severity level (that is, 0, 1, 2, 3, 4). Four of the items (irritability, speech, content, and disruptive-aggressive behavior) are scored 0 to 8 and have descriptors for every other increment (that is, 0, 2, 4, 6, 8). The item score is based on participant's report of his or her condition and clinician's behavioral observations during the interview, with emphasis on the latter. Higher scores indicate worsening. Responses are summed to yield YMRS total score ranging from 0 to 60.
Time Frame: Baseline and Endpoint (Week 13/LOCF) in OL Lead-in period, Endpoint (Week 25/LOCF) in open-label stabilization period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 667 | 0
Units on a scale
  OL Lead-in Period:Baseline (n=667) | 18.6 (9.48) |
  OL Lead-in Period:Change at Endpoint (n=653) | -9.9 (9.45) |
  OL Stabilization Period:Change at Endpoint (n=653) | -10.5 (10.14) |

11. Secondary Outcome: Double-blind: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Endpoint
Description: as for outcome 10
Time Frame: Baseline and Endpoint (Week 64/LOCF) in double-blind period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
Units on a scale
  Double-blind: Baseline (n=164, 170) | 4.4 (3.46) | 4.4 (3.40)
  Double-blind: Change at Endpoint (n=161,168) | -0.1 (5.47) | 3.2 (7.21)

12. Secondary Outcome: Open-label: Change From Baseline in Clinical Global Impression - Severity Schizoaffective Scale (CGI-S-SCA) Overall Score at Endpoint
Description: The CGI-S-SCA is a syndrome-specific 7-point scale (from 1 indicating not ill to 7 indicating very severely ill) that includes an overall severity score as well as scores for the positive, negative, manic, and depressive domains of the illness. The CGI-S-SCA was used to assess the level of overall impairment, as well as that related to each domain, at the time of the visit and for the week prior to the visit".
Time Frame: Baseline and Endpoint (Week 13/LOCF) in OL Lead-in period, Endpoint (Week 25/LOCF) in open-label stabilization period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 667 | 0
Units on a scale
  OL Lead-in Period:Baseline (n=667) | 4.4 (0.58) |
  OL Lead-in Period:Change at Endpoint (n=652) | -1.3 (0.99) |
  OL Stabilization Period:Change at Endpoint (n=652) | -1.3 (1.07) |

13. Secondary Outcome: Double-blind: Change From Baseline in Clinical Global Impression - Severity Schizoaffective Scale (CGI-S-SCA) Overall Score at Endpoint
Description: as for outcome 12
Time Frame: Baseline and Endpoint (Week 64/LOCF) in double-blind period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Placebo
Number analyzed (Participants) | 164 | 170
Units on a scale
  Double-blind: Baseline (n=164, 170) | 2.4 (0.68) | 2.5 (0.69)
  Double-blind: Change at Endpoint (n=161,168) | 0.0 (1.02) | 0.4 (1.15)

ADVERSE EVENTS:
Groups:
- Open Label - Paliperidone Palmitate: Open Label (OL) Lead-in (13 weeks): 234 milligram (mg) injection on Day 1, 156 mg on Day 8, flexible dose between 78-234 mg on Days 36, 64, and 92, given as monotherapy and as an adjunct to mood stabilizers or antidepressants. Participants who met criteria: Positive and Negative Syndrome Scale (PANSS) total score less than or equal to (<=) 70, and Young Mania Rating Scale [YMRS] and Hamilton Rating Scale for Depression [HAM-D-21] <=12 at the end of open label lead-in period entered stabilization period. OL Stabilization (12 weeks): Same dose as Day 92 in OL lead in period, on Day 120 once every 4 weeks, given as monotherapy and as an adjunct to mood stabilizers or antidepressants. Participants who completed stabilization period and maintained stabilization criteria throughout 12 weeks entered double- bind (DB) relapse prevention period.
- Double Blind - Paliperidone Palmitate: DB Relapse prevention period (15 months): Same dose as Day 92, once every 4 weeks, given as monotherapy and as an adjunct to mood stabilizers or antidepressants, until one of the following occurred: met the prospectively defined relapse criteria; discontinued treatment for a reason other than relapse; withdrew consent; lost to follow-up; completed 15 months of double-blind treatment.
- Double Blind - Placebo: Participants did not receive placebo during OL lead in period and OL stabilization period. Participants received matching placebo injections of 20 percent Intralipid (200 milligram per milliliter [mg/mL]) emulsion, once every 4 weeks, given as monotherapy and as an adjunct to mood stabilizers or antidepressants during DB relapse prevention period.
Arm/Group | Open Label - Paliperidone Palmitate | Double Blind - Paliperidone Palmitate | Double Blind - Placebo
Serious Adverse Events (participants affected / at risk) | 54/667 | 9/164 | 16/170
Other Adverse Events (participants affected / at risk) | 332/667 | 79/164 | 62/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label - Paliperidone Palmitate (N=667) | Double Blind - Paliperidone Palmitate (N=164) | Double Blind - Placebo (N=170)
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 1 | 0 | 0
Congestive Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Meniere's Disease (Ear and labyrinth disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 0
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Coma (Nervous system disorders) | 1 | 0 | 0
Viith Nerve Paralysis (Nervous system disorders) | 0 | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 2 | 0
Depression Suicidal (Psychiatric disorders) | 1 | 0 | 0
Depressive Symptom (Psychiatric disorders) | 2 | 0 | 0
Hallucination, Auditory (Psychiatric disorders) | 1 | 0 | 0
Homicidal Ideation (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 3 | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 4 | 2 | 2
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Schizoaffective Disorder (Psychiatric disorders) | 16 | 1 | 7
Suicidal Ideation (Psychiatric disorders) | 15 | 0 | 2
Suicide Attempt (Psychiatric disorders) | 2 | 0 | 0
Bladder Prolapse (Renal and urinary disorders) | 1 | 0 | 0
Therapy Regimen Changed (Surgical and medical procedures) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label - Paliperidone Palmitate (N=667) | Double Blind - Paliperidone Palmitate (N=164) | Double Blind - Placebo (N=170)
Hyperprolactinaemia (Endocrine disorders) | 9 | 7 | 2
Constipation (Gastrointestinal disorders) | 14 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 20 | 4 | 2
Dry Mouth (Gastrointestinal disorders) | 15 | 0 | 1
Nausea (Gastrointestinal disorders) | 17 | 2 | 3
Toothache (Gastrointestinal disorders) | 8 | 5 | 2
Fatigue (General disorders) | 20 | 3 | 0
Injection Site Pain (General disorders) | 71 | 1 | 2
Pyrexia (General disorders) | 8 | 6 | 2
Nasopharyngitis (Infections and infestations) | 9 | 9 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 14 | 7 | 4
Urinary Tract Infection (Infections and infestations) | 8 | 5 | 4
Blood Prolactin Increased (Investigations) | 4 | 4 | 2
Glycosylated Haemoglobin Increased (Investigations) | 1 | 2 | 4
Weight Decreased (Investigations) | 2 | 5 | 2
Weight Increased (Investigations) | 57 | 14 | 8
Increased Appetite (Metabolism and nutrition disorders) | 18 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 2 | 3
Akathisia (Nervous system disorders) | 74 | 5 | 3
Dyskinesia (Nervous system disorders) | 14 | 1 | 3
Headache (Nervous system disorders) | 36 | 9 | 6
Parkinsonism (Nervous system disorders) | 43 | 3 | 3
Somnolence (Nervous system disorders) | 21 | 2 | 2
Tremor (Nervous system disorders) | 23 | 2 | 4
Anxiety (Psychiatric disorders) | 9 | 3 | 4
Insomnia (Psychiatric disorders) | 67 | 8 | 12
Schizoaffective Disorder (Psychiatric disorders) | 6 | 4 | 3
Suicidal Ideation (Psychiatric disorders) | 16 | 5 | 2
Amenorrhoea (Reproductive system and breast disorders) | 18 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submitting a manuscript the Site shall provide to Sponsor a copy of all such manuscripts and materials,and allow Sponsor 60 days to review and comment on them. If Sponsor requests, the Site shall remove any Confidential Information prior to submitting the materials.The Site agrees that if Study is part of a multi-center study,any publication by the Institution of results of the Study conducted at the Site shall not be made before the first multi-center publication.